CLINICAL TRIAL: NCT04871958
Title: Individualized, Technological Interventions for Diabetes Care in the COVID-19 Ward
Acronym: Initiator
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Shift of the participating wards to non-Covid patients
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giovanni Annuzzi, Associate professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Initiator
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus; Covid19
Keywords: Diabetes mellitus; Covid-19; Hospital care; Continuous glucose monitoring; Insulin pump; CGM metrics
MeSH Terms: conditions — Diabetes Mellitus; COVID-19 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: All patients admitted at the COVID-19 non-ICU with a diagnosis of Type 2 or Secondary diabetes mellitus (DM) for whom intensive insulin therapy (basal plus at least two boluses) is indicated are eligible for the primary study.
  After stratification for admission ward, type of DM (known/unknown type 2, steroid use), age, and gender, participants will be randomized to one of the following interventions:
  1. Real-time CGM, multiple daily injections managed according to CGM
  2. Real-time CGM, insulin pump (V-Go) managed according to CGM
  3. Blind CGM, multiple daily injections managed according to POC glucose testing.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rtCGM/MDI (Experimental): Real-time CGM, insulin therapy by multiple daily injections managed according to CGM
  Interventions: Device: Continuous glucose monitoring (CGM, Dexcom G6)
- rtCGM/V-Go (Experimental): Real-time CGM, insulin therapy by V-Go insulin pump managed according to CGM
  Interventions: Device: Continuous glucose monitoring (CGM, Dexcom G6)
- blindCGM/MDI (No Intervention): Blind CGM, insulin therapy by multiple daily injections managed according to standard care (capillary glucose measurements)

INTERVENTIONS:
Device: Continuous glucose monitoring (CGM, Dexcom G6) — The Dexcom G6 sensor will be placed on the back of the upper arm at admission and changed after 10 days. In the participants randomized to Real-time CGM, glucose values will be transmitted through Bluetooth to a mobile phone at the bedside. From this phone data are transmitted to a tablet in the nursing station.
  In the blinded CGM group, sensor readings will be blinded to patient and healthcare providers.
  The MDI groups will be managed with basal/bolus insulin regimen, as clinically indicated.
  V-Go will be placed on the abdomen each morning. Insulin-naïve patients randomized to the V-Go system will start at the lowest basal rate (20 UI/24h).
  On daily basis, expert diabetologists will retrospectively review CGM data and provide indications for insulin therapy adjustments.
  Other Names: Continuous subcutaneous insulin infusion (V-Go)
  Arms: rtCGM/MDI; rtCGM/V-Go

SUMMARY:
During the current Covid-19 pandemic, many hospitals worldwide have been overwhelmed and strategies based on new technologies have been considered to improve the outcomes in patients with diabetes and Covid-19 and to prevent healthcare workers' exposure. Point-of-care blood glucose measurements, with the need of frequent and intermittent blood glucose testing and the associated time burden for hospital staff workers, have evident limitations. To this respect, continuous glucose monitoring (CGM) might represent an effective tool in hospitalized patients. The latest CGM devices have alarms alerting clinicians (or patients) to abnormal blood glucose values. Furthermore, CGMs not requiring calibration with capillary glucose testing have the potential to decrease both nurse and patient burden.

Insulin therapy is recommended in hospitalized patients with diabetes and Covid-19, conventionally by multiple daily insulin injections, i.e., rapid-acting insulin before meals and long-acting insulin once-a-day. Such a complex regimen demands also multiple daily fingerstick for glucose control. Use of continuous subcutaneous insulin infusion in hospital has been considered, and simple, less sophisticated pumps might be appro¬priate for prompt use by healthcare providers not specialized in diabetes treatment. V-Go® is a skin-patch insulin delivery device to be replaced every 24 h. It is fully mechanical, without tubing or electronics, and does not require any programming. It delivers a continuous basal infusion of rapid-acting insulin and allows for additional units before meals.

Therefore, the implementation of CGM and automated insulin infusion in Covid-19 hospitals has the potential to improve clinical outcomes, protect frontline healthcare workers, and preserve personal protective equipment. However, because only observational retrospective data for CGM use and no data on insulin pump use are currently available, randomized controlled trials are needed to determine whether using these technologies in hospital is of significant help.

The aims of this study are to explore, in patients with diabetes in COVID-19 wards, whether using continuous glucose monitoring with a glucose telemetry system and/or using a disposable insulin pump may improve blood glucose control and Covid-19 outcomes, and facilitate diabetes management.

DETAILED DESCRIPTION:
Both hyperglycaemia and hypoglycaemia are associated with poor outcomes in patients with COVID-19. In these patients, severe hyperglycaemia after hospital admission is a strong predictor of death among non-ICU patients and inpatient hyperglycaemia is associated with an increased risk of death even in patients without diabetes. However, there is no current indication for blood glucose targets in hospitalized patients with COVID-19.

During the current COVID-19 pandemic, many hospitals worldwide have been overwhelmed and diabetes care centers are considering strategies based on technology to improve the outcomes in patients with diabetes and COVID-19 and to prevent healthcare workers' exposure, while optimizing the use of personal protective equipment (PPE). Point-of-care (POC) blood glucose measurements, in the context of a Covid-19 ward, with the need of frequent and intermittent blood glucose testing and the associated time burden for nursing and ancillary hospital staff workers, have shown significant limitations. From this point of view, continuous glucose monitoring (CGM) might represent an effective tool for blood glucose tracking in hospitalized patients. Consistently, in April 2020 the FDA authorized the use of CGM in patients with Covid-19, making CGM a potential favoured option in these patients. Companies, like Abbott and Dexcom, have supplied CGM systems to hospitals and provided education to use their devices effectively. The latest generation of CGM devices have alarms that can alert clinicians (or patients) to abnormal blood glucose values. Furthermore, CGMs that no longer require calibration with POC glucose testing (factory-calibrated) have the potential to decrease both nurse and patient burden associated with frequent POC glucose testing in the hospital.

Healthcare professional societies recommend insulin therapy in hospitalized patients with diabetes, and this holds especially true in Covid-19 patients. The conventional treatment approach involves multiple daily insulin injections (MDI) and includes the administration of rapid-acting insulin analogues before meals and a long-acting insulin analogue once a day. Such a complex regimen demands also multiple daily POC fingerstick for glucose control. Automated insulin delivery including CSII (continuous subcutaneous insulin infusion) has been considered in the hospital setting. In type 2 diabetes, insulin pump therapy induces better glycaemic control than MDI. A likely mechanism for the improved control on CSII is that the traditional large bolus injections of long-acting insulin required during MDI in type 2 diabetes are more erratically absorbed than the slow rapid-acting insulin infusion of CSII. In this respect, the same dose of insulin given via the basal rate of CSII induced better glycaemic control and higher circulating serum insulin concentrations than when given as an injection of long-acting insulin.

However, starting and managing CSII in the hospital setting by personnel and patients not adequately trained might represent a challenging barrier in a Covid-19 ward. Therefore, simpler and less sophisticated pumps might become more appropriate for prompt use by healthcare providers not specialized in diabetes treatment. V-Go® (Zealand Pharma A/S, Denmark) is a wearable insulin delivery device, fully mechanical without tubing or electronics, that does not require any programming. It delivers a continuous basal infusion of rapid-acting insulin (20, 30, or 40 units/24 h) and allows for up to 36 additional units for mealtime dosing in 2-unit increments. V-Go® is filled with fast-acting insulin and is worn like a patch on the skin using a hypoallergenic and latex-free adhesive. It is designed to be replaced every 24 h and is fully disposable. The implant of the device is easily obtained by the push of a button that inserts a 4.6-mm, 30-gauge stainless steel needle subcutaneously and starts the delivery of the continuous pre-set basal rate of insulin. Mealtime bolus insulin doses are administered on-demand by pressing the bolus-ready button and the bolus delivery button. Previous studies showed that switching patients from traditional insulin delivery modes to V-Go® was associated with significantly improved glycaemic control.

Therefore, the implementation of CGM and insulin infusion technologies in Covid-19 hospitals has the potential to improve clinical outcomes, help to protect frontline healthcare workers, and preserve PPE. However, because only observational retrospective data for CGM use and no data on insulin pump use are currently available, randomized controlled trials are needed to determine whether use of CGM and CSII systems in the hospital can be of significant help.

The aims of this study are to explore whether in patients hospitalized in COVID-19 non-ICU:

1. the use of CGM with a glucose telemetry system, compared with intermittent capillary blood glucose monitoring and/or
2. the use of a disposable insulin pump, compared with a conventional multiple daily insulin injection, may improve blood glucose control and COVID outcomes in patients with type 2 or secondary diabetes mellitus and facilitate diabetes management by health care providers.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted at the COVID-19 non-ICU with a diagnosis of Type 2 or Secondary diabetes mellitus (DM) for whom intensive insulin therapy (basal plus at least two boluses) is indicated are eligible for the study.

Exclusion Criteria:

* Patients on hydroxyurea treatment are excluded (interference with glucose sensor readings).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Blood glucose Time-In-Range (TIR) during hospital stay | From date of randomization until the date of discharge from the hospital ward up to 2 months
  Percentage of time spent within the interval of blood glucose between 70 and 180 mg/dl

SECONDARY OUTCOMES:
Hypoglycemia events | From date of randomization until the date of discharge from the hospital ward up to 2 months
  Number and duration of hypoglycemias
Change in fructosamine | Date of admission and day of discharge from the hospital ward
  Change in fructosamine level during hospital stay
Change in COVID-19 severity score | Date of admission and day of discharge from the hospital ward
  Scores MEWS and SCARP
Length of stay in the hospital ward | From date of randomization until the date of discharge from the hospital ward up to 2 months
  Duration of stay
Accesses to the isolation room | From date of randomization until the date of discharge from the hospital ward up to 2 months
  Number of healthcare workers accesses to the isolation room (capillary blood glucose, insulin injections, other)

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University Hospital, Naples, Italy